CLINICAL TRIAL: NCT07069205
Title: "The Effect of Breathing Exercise Education and Follow-Up Supported by Tele-Nursing on Dyspnea and Quality of Life in Patients With Tuberculosis: A Single-Group Experimental Study"
Brief Title: Breathing Exercise and Tele-Nursing Support for Patients With Tuberculosis: A Single-Group Experimental Study
Acronym: TELEBREATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canan Güngör (Other)
Responsible Party: Sponsor-Investigator, Canan Güngör, PhD student, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: GUNGOR2025-TELEHEM; "03-663" (Other: Ankara Yıldırım Beyazıt Üniversitesi Sağlık Bilimleri Enstitüsü Etik Kurulu)
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Impaired Quality of Life; Pulmonary Tuberculosis (TB)
Keywords: Tele-nursing; Dyspnea; Quality of life; Telehealth
MeSH Terms: conditions — Tuberculosis, Pulmonary; Dyspnea

STUDY DESIGN:
Intervention Model Description: This study was conducted using a single-group pretest-posttest quasi-experimental design. All participants received the same structured respiratory exercise training and tele-nursing follow-up for 12 weeks.
Masking Description: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants receive tele-nursing supported respiratory exercises including abdominal breathing, pursed-lip breathing, and effective coughing training supported by educational booklets and videos over a 12-week period.
  Interventions: Behavioral: Tele-nursing supported respiratory exercises

INTERVENTIONS:
Behavioral: Tele-nursing supported respiratory exercises — This intervention consists of a structured tele-nursing supported respiratory exercise program including abdominal breathing, pursed-lip breathing, and effective coughing techniques. The training is delivered through educational booklets and videos over a 12-week period, aiming to improve respiratory function and patient self-management in tuberculosis patients.

SUMMARY:
This study was conducted as a single-group, pretest-posttest quasi-experimental design. The sample consisted of 54 tuberculosis patients registered at a Tuberculosis Dispensary who met the inclusion criteria and agreed to participate. Data collection tools included the Patient Identification Form, Dyspnea-12 TR Scale, Multidimensional Quality of Life Scale (MILQ), London Chest Activities of Daily Living Scale (LCADL), Tele-Nursing Follow-up Form, and Tele-Nursing Evaluation Form. Descriptive statistics, paired sample t-test, and Wilcoxon Signed-Rank Test were used for data analysis. The intervention group received structured respiratory exercises training, including abdominal breathing, pursed-lip breathing, and effective coughing, through educational materials (booklet and videos) developed by the researcher. Patients were regularly monitored for 12 weeks via phone calls and video conferencing. Baseline assessments were conducted using data collection tools at the first visit, and post-intervention assessments were performed at the end of week 12 to evaluate the effectiveness of the intervention.

DETAILED DESCRIPTION:
This study implemented a structured respiratory exercise intervention supported by tele-nursing to assess its impact on dyspnea severity and quality of life among patients diagnosed with tuberculosis. The intervention included abdominal breathing, pursed-lip breathing, and effective coughing techniques delivered through a combination of printed educational booklets and instructional videos. These materials were specifically developed for the study and validated by expert healthcare professionals to ensure content accuracy and cultural appropriateness.

Patients were monitored remotely over a 12-week period with scheduled weekly follow-up sessions conducted via telephone and video calls. These sessions facilitated reinforcement of the respiratory exercises, addressed patient inquiries, and enabled continuous assessment of adherence and response to the intervention. Data collection instruments, including validated Turkish versions of the Dyspnea-12 scale, the Multidimensional Quality of Life Scale (MILQ), and the London Chest Activities of Daily Living Scale (LCADL), were employed to quantitatively measure changes in respiratory symptoms, functional capacity, and overall quality of life.

Comprehensive data management protocols were followed to ensure confidentiality and data integrity throughout the study period. Statistical analyses were performed using appropriate parametric and non-parametric tests based on data distribution, including paired-sample t-tests and Wilcoxon Signed-Rank tests, to evaluate the pre- and post-intervention effects.

Ethical approval was obtained from the relevant institutional review board, and all participants provided informed consent prior to inclusion. This research contributes valuable insights into the feasibility and effectiveness of telehealth-supported respiratory therapy interventions in tuberculosis care, highlighting the potential of patient-centered, remotely delivered nursing practices to enhance treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with tuberculosis and registered at a Tuberculosis Dispensary.

Meets criteria for study participation.

Provides informed consent.

Able to participate in tele-nursing supported respiratory exercises and follow-up.

Exclusion Criteria:

Severe respiratory comorbidities preventing exercise participation.

Cognitive or communication impairments interfering with tele-nursing.

Declines to participate or unable to comply with intervention protocol.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Dyspnea Severity Using the Dispne-12 Turkish Version Scale | Baseline and at 12 weeks post-intervention
  This outcome measures the change in dyspnea severity in tuberculosis patients before and after receiving tele-nursing supported respiratory exercise training over 12 weeks, using the validated Dispne-12 TR scale.
Change in Dyspnea Severity (Dispne-12 TR Scale) | Baseline (pre-intervention) and 12 weeks after the intervention.
  The change in dyspnea severity will be measured using the Dispne-12 Turkish version scale to assess the effectiveness of tele-nursing supported respiratory exercises on patients with tuberculosis over a 12-week period.

CONTACTS AND LOCATIONS:
Overall Officials: Canan Güngör, RN, Study Chair — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yıldırım Beyazıt Üniversitesi Sağlık Bilimleri Enstitüsü, Ankara, Ankara, Turkey (Türkiye)